CLINICAL TRIAL: NCT02550782
Title: Does Patient-Controlled Infraclavicular Perineural Dexmedetomidine Improve Postoperative Analgesia Deadline?
Brief Title: Infraclavicular Perineural Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, Anaesthesiology and reanimation, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Mengücek gazi
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: The Analgesic Effects
Keywords: perineural dexmedetomidine; infraclavicular perineural catheter; postoperative analgesia
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- perineural bupivacaine (Active Comparator): patient-controlled infraclavicular perineural bupivacaine
  (1% bupivacaine (marcaine), 5 ml bolus dose, infusion rate of 5 ml / h, lockout time 1 hour)
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine
- perineural dexmedetomidine (Experimental): patient-controlled infraclavicular perineural dexmedetomidine
  (1% bupivacaine + 200 mic / 100cc dexmedetomidine, 5 ml bolus dose, infusion rate of 5 ml / h, lockout time 1 hour)
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — patient- controlled infraclavicular perineural marcaine infusion
Drug: Dexmedetomidine — patient- controlled infraclavicular perineural marcaine with dexmedetomidine infusion

SUMMARY:
Infraclavicular block is one of the peripheral nerve block used in upper extremity surgery. Adjuvant agents are used in peripheral nerve blocks to increase the duration and block quality. We investigated that the effects of patient-controlled perineural dexmedetomidine application on postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* be undergoing distal upper extremity surgery
* Be between 18-65 years
* to agree to participate in research

Exclusion Criteria:

* allergy to dexmedetomidine
* AV block or bradycardia
* being serious cardiac - liver - kidney function disorders
* Being coagulopathy
* neuropathy in the upper extremity
* adrenoceptor agonists or antagonists use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 3 month
  Scores range from 0 [no pain] to 10 [worst possible pain

SECONDARY OUTCOMES:
side effects | 3 month
The effect of dexmedetomidine to the Ramsey Sedation Scale | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Üniversity, Erzincan, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Latifzai K, Sites BD, Koval KJ. Orthopaedic anesthesia - part 2. Common techniques of regional anesthesia in orthopaedics. Bull NYU Hosp Jt Dis. 2008;66(4):306-16. PMID 19093908
- [Background] Mariano ER, Loland VJ, Sandhu NS, Bishop ML, Lee DK, Schwartz AK, Girard PJ, Ferguson EJ, Ilfeld BM. Comparative efficacy of ultrasound-guided and stimulating popliteal-sciatic perineural catheters for postoperative analgesia. Can J Anaesth. 2010 Oct;57(10):919-26. doi: 10.1007/s12630-010-9364-7. Epub 2010 Aug 11. PMID 20700680
- [Background] Gray AT, Collins AB, Schafhalter-Zoppoth I. An introduction to femoral nerve and associated lumbar plexus nerve blocks under ultrasonic guidance. Tech Reg Ananesth Pain Man. 2004;8:155-63.
- [Background] Greengrass R, Steele S, Moretti G. Peripheral nerve blocks. In: Raj PP, editor. Textbook of regional anesthesia. New York: Churchill Livingstone; 2002. p. 325-77.
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] di Benedetto P, Casati A, Bertini L, Fanelli G, Chelly JE. Postoperative analgesia with continuous sciatic nerve block after foot surgery: a prospective, randomized comparison between the popliteal and subgluteal approaches. Anesth Analg. 2002 Apr;94(4):996-1000, table of contents. doi: 10.1097/00000539-200204000-00041. PMID 11916811
- [Result] Svediene S, Andrijauskas A, Ivaskevicius J, Saikus A. The efficacy comparison of on-demand boluses with and without basal infusion of 0.1 % bupivacaine via perineural femoral catheter after arthroscopic ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2013 Mar;21(3):641-5. doi: 10.1007/s00167-012-1971-0. Epub 2012 Apr 13. PMID 22527409
- [Result] Song JH, Shim HY, Lee TJ, Jung JK, Cha YD, Lee DI, Kim GW, Han JU. Comparison of dexmedetomidine and epinephrine as an adjuvant to 1% mepivacaine in brachial plexus block. Korean J Anesthesiol. 2014 Apr;66(4):283-9. doi: 10.4097/kjae.2014.66.4.283. Epub 2014 Apr 28. PMID 24851163